CLINICAL TRIAL: NCT02312661
Title: Phase Ib Study of Metformin in Combination With Carboplatin/Paclitaxel Chemotherapy in Patients With Advanced Ovarian Cancer
Brief Title: Study of Metformin With Carboplatin/Paclitaxel Chemotherapy in Patients With Advanced Ovarian Cancer
Acronym: OVMET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30102012
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Epithelial Ovarian Cancer
Keywords: ovarian cancer; metformin; carboplatin; paclitaxel
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Metformin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin / paclitaxel /metformin (Experimental): Three-weekly cycles of carboplatin/paclitaxel chemotherapy in combination with metformin treatment
  Interventions: Drug: Metformin; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Metformin — Metformin in increasing doses will be added to carboplatin/paclitaxel chemotherapy
Drug: Carboplatin — Intravenous carboplatin chemotherapy in three-weekly cycles, for a maximum of 6 cycles
Drug: Paclitaxel — Intravenous paclitaxel chemotherapy in three-weekly cycles, for a maximum of 6 cycles

SUMMARY:
Molecularly targeted agents which inhibit the mammalian target of rapamycin (mTOR) pathway and/or circumvent p53 in the induction of apoptosis are exciting potential targets in ovarian cancer. Metformin is a biguanide, widely used in the treatment of type 2 diabetes mellitus, that has shown anti-cancer activity in preclinical studies. The main mechanism of metformin's effect is mTOR pathway inhibition and, in addition, it has been shown to circumvent p53-induced apoptosis making it an exciting, potentially effective drug in ovarian cancer.

DETAILED DESCRIPTION:
A phase Ib, single-centre, dose-escalation trial with a traditional escalation rule with fixed dose levels ("3 + 3" rule). The recommended phase II dose will be defined as the maximum predefined dose level at which 0 of 3 or ≤ 1 of 6 subjects experience a drug-related dose limiting toxicity (DLT) during cycle 1 and 2 of treatment. An estimated 10-20 patients will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage (FIGO III-IV), histologically confirmed and documented epithelial ovarian carcinoma
* Patients eligible for neo-adjuvant carboplatin/paclitaxel chemotherapy prior to surgical debulking OR patients with relapsed or progressive ovarian cancer after initial treatment eligible for palliative carboplatin/paclitaxel chemotherapy
* Eastern Cooperative Oncology Group-performance status (ECOG-PS) of 0-2
* Age ≥ 18 years
* Laboratory Requirements - within 7 days prior to enrolment:
* absolute neutrophil count (ANC) ≥1.5 x 109/L
* platelets > 100 x 109/L
* hemoglobin >9g/dl. Patients may be transfused or use erythropoietin to maintain hemoglobin values ≥ 9 g/dl.
* hepatic function: bilirubin ≤1.5×upper limit of normal (ULN), aspartate aminotransferase (AST)/ALT≤2.5×ULN
* estimated creatinine clearance ≥ 60ml/min
* Before patient registration/randomization, written informed consent for the trial must be given according to International Conference on Harmonisation (ICH)/ good clinical practice (GCP), and national/local regulations.

Exclusion Criteria:

* Current or recent (within 30 days of first study dosing) treatment with another investigational drug or participation in another investigational study.
* Metformin within 4 weeks prior to enrolment.
* Symptomatic central nervous system (CNS) metastasis
* Pre-existing peripheral neuropathy ≥ Common toxicity criteria (CTC) grade 2.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start.
* Women of childbearing potential (defined as <2 years after last menstruation and not surgically sterile) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly) during the study and for 6 months after the last study medication.
* Known hypersensitivity to any of the study drugs or excipients.
* Serious active infection requiring i.v. antibiotics at enrolment.
* Unstable medical conditions.
* Evidence of any other medical conditions, physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a measure of safety and tolerability | 1-2 years
  Data will be used to determine recommended phase 2 dose

SECONDARY OUTCOMES:
Pharmacokinetics (AUC, Tmax,Cmax) of carboplatin and paclitaxel chemotherapie | 1-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Mecdical Center Groningen, Groningen, Netherlands